CLINICAL TRIAL: NCT02590939
Title: Multi-center, Double-blind, Randomized, Sham-controlled Trial on the Acute Treatment of Migraine With the Cefaly® Device
Brief Title: Acute Treatment of Migraine With e-TNS
Acronym: ACME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 50213
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active device (Experimental): 60 minutes of active external trigeminal nerve stimulation with a CEFALY Active device
  Interventions: Device: CEFALY Active
- Sham device (Sham Comparator): 60 minutes of placebo external trigeminal nerve stimulation with a CEFALY Placebo device
  Interventions: Device: CEFALY Placebo

INTERVENTIONS:
Device: CEFALY Active — Active external trigeminal nerve stimulation
  Arms: Active device
Device: CEFALY Placebo — Placebo external trigeminal nerve stimulation
  Arms: Sham device

SUMMARY:
The main objective of this study is to assess the efficacy of the Cefaly® device as an acute treatment of migraine attack in adult patients. The patients will be applied either an active or placebo external neurostimulation for 1 hour during a migraine attack, and will report the pain on a visual analog scale before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of episodic or chronic migraine with or without aura meeting the diagnostic criteria listed in ICHD-III beta (2013) section 1, migraine, with the exception of ''complicated migraine'' (i.e., hemiplegic migraine, basilar-type migraine, ophthalmoplegic migraine, migrainous infarction)
* Having a migraine attack lasting at least 3 hours
* Migraine pain intensity stabilized for at least 1 hour
* Frontal, retro-, or peri- orbital headache.

Exclusion Criteria:

* Pregnant women
* Patients having received Botox treatment in the prior 4 months
* Patients having received supraorbital nerve blocks in the prior 4 months
* Diagnosis of other primary or secondary headache disorders, except of Medication Overuse Headache
* Patients with only temporal or occipital headache
* Patients using opioid medication
* Patients having taken abortive migraine medication in the prior 3 hours
* Allodynia: intolerance to supraorbital neurostimulation (allodynia) that makes the treatment not applicable (the patients will be excluded if they are unable to tolerate the first 5 minutes of neurostimulation).
* Implanted metal or electrical devices in the head
* Cardiac pacemaker or implanted or wearable defibrillator
* Patient having had a previous experience with Cefaly®

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Chou, M.D., Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Rowe Neurology Institute, Lenexa, Kansas
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Derived] Chou DE, Shnayderman Yugrakh M, Winegarner D, Rowe V, Kuruvilla D, Schoenen J. Acute migraine therapy with external trigeminal neurostimulation (ACME): A randomized controlled trial. Cephalalgia. 2019 Jan;39(1):3-14. doi: 10.1177/0333102418811573. Epub 2018 Nov 17. PMID 30449151

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Device: 60 minutes of active external trigeminal nerve stimulation with a CEFALY device
  CEFALY Active: Active external trigeminal nerve stimulation
- Sham Device: 60 minutes of placebo external trigeminal nerve stimulation with a CEFALY device
  CEFALY Placebo: Placebo external trigeminal nerve stimulation
Period: Overall Study
Arm/Group | Active Device | Sham Device
Started | 52 | 54
Completed | 47 | 52
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Failed the nociceptive test | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Device | Sham Device | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.71 (13.62) | 40.09 (12.65) | 39.90 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 49 | 92
  Male | 9 | 5 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Migraine type [Count of Participants; unit: Participants]
  Migraine with aura | 12 | 5 | 17
  Migraine without aura | 40 | 49 | 89
Migraine duration (hours) [Median (Inter-Quartile Range); unit: hours] | 7 [4 to 48] | 6 [4.63 to 20.75] | 6 [4 to 24]
Use of acute medication before enrollment [Count of Participants; unit: Participants] | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Pain Score 1-hour
Description: Mean change of pain score (measured on a pain visual analog scale containing 11 values, from 0 to 10, with 0 meaning no pain and 10 meaning maximal pain) at 1 hour compared to baseline
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
percent change | -59 (35) | -30 (31)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pain Score 1-hour
Description: as for outcome 1
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
units on a scale | -3.46 (2.32) | -1.78 (1.89)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Rescue Medication 2 Hours
Description: Number of patients not having required rescue medication at 2 hours
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
Participants
  Patients having used rescue medication at 2 hours | 3 | 2
  Patients not having used rescue medication at 2 h | 44 | 50
  Patients for whom med data was not available | 5 | 2
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p = 0.666, Fisher Exact — Statistical significance threshold set to 0.05

4. Secondary Outcome: Pain Score 2 Hours
Description: Mean change of pain score (measured on a pain visual analog scale containing 11 values, from 0 to 10, with 0 meaning no pain and 10 meaning maximal pain) at 2 hours compared to baseline (if rescue therapy was not used)
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
percent change | -50 (36) | -32 (37)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p = 0.026, Wilcoxon (Mann-Whitney) — Statistical significance threshold set to 0.05

5. Secondary Outcome: Rescue Medication 24 Hours
Description: Number of patients not having required rescue medication within 24 hours
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
Participants
  Patients having used rescue medication within 24 h | 18 | 21
  Patients not having used rescue med within 24h | 27 | 30
  Patients for whom med data was not available | 7 | 3
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney) — Statistical significance threshold set to 0.05

6. Secondary Outcome: Pain Score 24 Hours
Description: Mean change of pain score (measured on a pain visual analog scale containing 11 values, from 0 to 10, with 0 meaning no pain and 10 meaning maximal pain) at 24 hours compared to baseline (if rescue therapy was not used)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
percent change | -57 (37) | -40 (40)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p = 0.037, Wilcoxon (Mann-Whitney) — Statistical significance threshold set to 0.05

7. Secondary Outcome: Pain Score 2 Hours
Description: as for outcome 4
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
units on a scale | -2.87 (2.24) | -1.85 (1.96)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney) — Statistical significance threshold set to 0.05

8. Secondary Outcome: Pain Score 24 Hours
Description: as for outcome 6
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 52 | 54
units on a scale | -3.46 (2.65) | -2.38 (2.27)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Test type: Superiority; p = 0.062, Wilcoxon (Mann-Whitney) — Statistical significance threshold set to 0.05

ADVERSE EVENTS:
Time Frame: 24 hours following the beginning of the treatment
Arm/Group | Active Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54
Other Adverse Events (participants affected / at risk) | 1/52 | 0/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Device (N=52) | Sham Device (N=54)
Nausea (Nervous system disorders) | 1 (1) | 0 (0) — After ending the session early (7 minutes), the patient reported nausea that was not present prior to treatment; the nausea resolved without intervention after 20 minutes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 60 days from the time submitted to the sponsor for review. Sponsor may request:

* deletion of any trade secret, proprietary, or confidential information of Sponsor
* an additional 90 days to take measures to preserve its IP rights

Sponsor cannot require editorial changes. Sponsor's consent is required for results communication before trial completion

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT02590939/Prot_SAP_000.pdf